CLINICAL TRIAL: NCT05376280
Title: Nutritional Assessment in Non-tuberculous Mycobacteria Pulmonary Disease: an Exploratory Study
Brief Title: Nutritional Assessment in Non-tuberculous Mycobacteria Pulmonary Disease
Acronym: nutriNTM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Paola Faverio, Doctor, University of Milano Bicocca
Other Study IDs: nutriNTM
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Non-Tuberculous Mycobacterial Pneumonia
Keywords: nutrition; nutritional status; sarcopenia; malnutrition; body mass index; bioimpedance analysis
MeSH Terms: conditions — Sarcopenia; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-tuberculous mycobacterial (NTM) pulmonary disease (PD) is an emerging condition with heterogeneous manifestations from both the microbiological and the clinical point of view. Diagnostic and therapeutic guidelines are available but there are still unmet patients' and physicians' needs, including the exams to perform in the nutritional evaluation and intervention to improve health-related QoL and to control gastrointestinal side-effects during antimicrobial therapy, particularly in those with low body mass index and history of weight loss.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the nutritional status in patients with non-tuberculous mycobacterial pulmonary disease (NTM-PD) and to provide an initial assessment of the potential impact of the introduction of targeted antibiotic therapy on the nutritional status itself.

Specifically, the primary objective is the assessment of the proportion of underweight subjects, i.e. with Body Mass Index (BMI) <18.5 kg/m2, to confirm that it is significantly higher than that of the general Italian population.

Study Design: Multicenter Cohort Pilot Observational Study

Participation in the study consists of two pneumological visits, as per normal clinical practice, (at the beginning of the study, T1, after 6 months, T3, and at the end of the antimicobacterial antibiotic therapy, T5) in which the collection of past medical history, measurement of oxygen saturation, pulmonary functional tests and 6-minute walking tests will be performed. In addition, nutritional assessments (T2, T4, T6) will be carried out at the same time as the pulmonary visits. Nutritional assessments will include anthropometric measurements, questionnaires on nutritional status and physical activity, performing blood chemistry tests, bioimpedance, dynamometry and gait speed 4 meters, to evaluate body composition and physical performance.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18 years;
* diagnosis of NTM-PD according to the BTS 2017 guidelines

Exclusion Criteria:

* severe renal failure, defined as a GFR (glomerular filtration rate) lower than 30ml / min; NYHA class IV;
* severe liver failure, defined as Child-Pugh score class C;
* active solid or haematological neoplasms;
* having already received (currently or in the prior 6 months) antimicobacterial therapy;
* severe immunosuppression;
* inability to walk without help;
* need for oxygen therapy at rest;
* participation in other interventional experimental protocols with use of a medicinal product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a recent diagnosis of NTM-PD
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
BMI (body mass index) | baseline (NTM-PD diagnosis)
  kg/m2

SECONDARY OUTCOMES:
FFMI (fat free mass index) | baseline (NTM-PD diagnosis), 6-month follow-up, 12-month follow-up
  kg/m2
SMI (skeletal muscle mass index) | baseline (NTM-PD diagnosis), 6-month follow-up, 12-month follow-up
  kg/m2
BFMI (body fat mass index) | baseline (NTM-PD diagnosis), 6-month follow-up, 12-month follow-up
  kg/m2
Hand grip | baseline (NTM-PD diagnosis), 6-month follow-up, 12-month follow-up
  kg/m2
Abdominal circumference | baseline (NTM-PD diagnosis), 6-month follow-up, 12-month follow-up
  cm
Malnutrition Universal Screening Tool (MUST) Screening Tool (MUST) | baseline (NTM-PD diagnosis), 6-month follow-up, 12-month follow-up
  questionnaire score: score 0 = low risk of malnutrition; score 1 = medium risk of malnutrition; score equal or higher than 2 = high risk of malnutrition
Mini Nutritional Assessment (MNA) | baseline (NTM-PD diagnosis), 6-month follow-up, 12-month follow-up
  questionnaire score (maximum score 30): total score > 23.5 = normal nutritional status; total score < 23.5 = inadequate nutritional status
plasma vitamin D | baseline (NTM-PD diagnosis), 6-month follow-up, 12-month follow-up
  vitamin D level in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Gerardo dei Tintori, Monza, MB, Italy